CLINICAL TRIAL: NCT05180994
Title: Topical Infliximab in Eyes With Penetrating Keratoplasty
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de recherche en ophtalmologie de l'Université de Montréal (Other); Maisonneuve-Rosemont Hospital (Other); Niagara Health System (Other); Prism Eye Institute (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CE 21.232; MP-02-2021-9824 (Other: Centre Hospitalier de l'Université de Montréal)
Record Dates: First submitted 2021-11-29; First posted 2022-01-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma Following Surgery
MeSH Terms: interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical infliximab following PKP surgery (Experimental): Additionally to standard post-operative regimen, patients who will be undergoing their first PKP surgery and who meet all inclusion and no exclusion criteria will be included in the experimental group. These patients will administer topical infliximab four times per day for 3 months.
  Interventions: Drug: Topical infliximab
- No topical infliximab following PKP surgery (Active Comparator): Patients who will be undergoing their first PKP surgery, but who are not qualified to receive infliximab or who refuse to receive infliximab, will be included in the control group. These patients will only administer the standard post-operative regimen following their PKP surgery and will not administer topical infliximab. They will be followed with the same follow-up schedule, questionnaires, examinations and non-invasive tests (excluding lab work) as patients in the interventional group.
  Interventions: Other: No topical infliximab

INTERVENTIONS:
Drug: Topical infliximab — Infliximab eye drops (10mg/ml) administered four (4) times per day for three (3) months.
  Other Names: Remicade
  Arms: Topical infliximab following PKP surgery
Other: No topical infliximab — No treatment with infliximab.
  Arms: No topical infliximab following PKP surgery

SUMMARY:
Penetrating keratoplasty is a cornea surgery involving several inflammatory complications, of which the most important is glaucoma. Researchers wish to determine whether it is safe to administer infliximab (an anti-inflammatory drug) eye drops after surgery, and whether this eye drop could prevent the occurrence of glaucoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, double-arm open clinical trial of 50 patients receiving a first penetrating keratoplasty (PKP) surgery, recruited to receive infliximab drops post-operatively.

The current study aims to evaluate whether using topical infliximab 10mg/ml eye drops is safe and efficient to prevent the emergence of glaucoma of inflammatory etiology in patients with PKP. This study is examining a new form of delivering infliximab (as eye drops instead of injections in the veins). 25 patients who will be undergoing PKP surgery will be recruited to receive infliximab drops as a part of this study.

The research hypothesis is that topical infliximab used during the PKP post-operative period will be safe, and could protect against the occurrence of glaucoma.

For comparison purposes, if some patients are not qualified to receive infliximab or should they refuse to receive infliximab, these patients will still be offered to follow the same follow-up schedule, questionnaires, examinations and non-invasive tests (excluding lab work), as patients who will be receiving infliximab. The number of patients in this control group will also be limited to 25 patients.

During the treatment period, patients in the interventional arm of the study will be receiving topical infliximab 10mg/ml eye drops four times per day, for a duration of 3 months. Patients will be monitored for another 3 months after cessation of the study drug. The total study duration for each patient will be 6 months.

Regarding statistical analysis, the primary and secondary outcomes of the study will be described, including : percentage of patients presenting with a thinning of mean retinal nerve fiber thickness measured using OCT (optical coherence tomography), with thinning in four quadrants (inferior, superior, nasal, temporal); proportion of patients without glaucoma over time; mean change in BCVA (best corrected visual acuity) compared to baseline BCVA; OSDI (Ocular Surface Disease Index) score evolution over time; quantification of ocular surface inflammation; quantification of anterior chamber inflammation; epithelial healing time; and incidence of epithelial keratitis.

Visual acuity values will be converted to LogMAR. Data will be presented as numbers and percentages for categorical variables, and as mean ± standard deviation for continuous variables. Comparison between experimental and comparison groups will be done using student's t test if distribution is parametric, and Mann-Whitney U test if distribution is non-parametric. The Kaplan-Meier curve will be used in order to illustrate the proportion of patients without glaucoma over time. An interim statistical analysis will be done once n=10 patients will have completed the full 6 months of study follow-up. A statistical significance level of α=0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* First corneal transplant surgery;
* Capable of providing informed consent;
* Capable of administering eye medication or access to a caregiver able and willing to administer the eye medication for the patient.

Exclusion Criteria:

* Active ocular infection;
* Past corneal transplant (any technique);
* Advanced glaucoma or macular disease;
* Active or latent systemic infection (tuberculosis, histoplasmosis, coccidioidomycosis, cytomegalovirus, pneumocystis, aspergillosis or hepatitis B);
* Malignancy diagnosed in the past 5 years (any kind);
* Demyelinating disease;
* History or current diabetes mellitus (controlled or uncontrolled) or heart failure (New York Heart Association class III or IV);
* Pregnancy or breastfeeding;
* Allergy to infliximab or to a compound of its topical formulation;
* Significant anomaly of complete blood count or hepatic enzymes;
* Current or anterior use of anti-TNF-α medication or other anti-inflammatory biologics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Complications associated to PKP surgery | 6 months
  Number and type of complications associated to PKP surgery (graft loss, infectious keratitis, graft failure, corneal melting…)
Complications associated to infliximab use | 6 months
  Number and type of complications associated with infliximab use (serious infections, allergic reactions, heart failure, blood problems, nervous system disorders, malignancies…; these complications have been observed with intravenous infliximab administration).

SECONDARY OUTCOMES:
Mean retinal nerve fiber thickness | 6 months
  Percentage of patients presenting with a thinning of mean retinal nerve fiber thickness measured using OCT, with thinning in four quadrants (inferior, superior, nasal, temporal).
Occurrence of glaucoma | 6 months
  Proportion of patients without glaucoma over time.
Best Corrected Visual Acuity (BCVA) | 6 months
  Mean change in BCVA compared to baseline BCVA, measured using a Snellen chart.
Ocular surface symptoms | 6 months
  Ocular surface symptoms as assessed by the Ocular Surface Disease Index (OSDI) questionnaire, ranging from 0 to 100, where a higher score indicates increased disease severity.
Quantification of ocular surface inflammation | 6 months
  Conjunctival erythema on a scale of 0 to 4, where a higher score indicates increased disease severity.
Quantification of anterior chamber inflammation | 6 months
  Quantification of anterior chamber inflammation according to the SUN definition (Standardization of Uveitis Nomenclature).
Epithelial healing time | 6 months
  Number of days between surgery and absence of epithelial deficit.
Incidence of epithelial keratitis | 6 months
  Incidence of epithelial keratitis assessed using the National Eye Institute Score (0-15).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Robert, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No